CLINICAL TRIAL: NCT00779389
Title: Comparison of Biomarker Modulation by Inhibition of EGFR and/or Src Family Kinases Using Erlotinib and Dasatinib in Head and Neck Lung Cancers
Brief Title: Comparison of Biomarker Modulation by Inhibition of EGFR and/or SRC Family
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-124
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-02

CONDITIONS: Head and Neck Cancer; Non Small Cell Lung Cancer
Keywords: Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Dasatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental): Erlotinib 150 mg
  Interventions: Drug: Erlotinib
- Arm B (Experimental): Dasatinib + placebo
  Interventions: Drug: Dasatinib + Placebo
- Arm C (Experimental): Erlotinib (150 mg) plus Dasatinib (100 mg) for 14-21 days.
  Interventions: Drug: Erlotinib plus Dasatinib
- Arm D (Placebo Comparator): Placebo for 14-21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150mg will be taken once a day for 14-21days.
  Other Names: Tarceva
  Arms: Arm A
Drug: Dasatinib + Placebo — Dasatinib (100 mg) once a day for 14-21 days.
  Other Names: Sprycel
  Arms: Arm B
Drug: Erlotinib plus Dasatinib — Erlotinib (150 mg PO qD) plus Dasatinib (100 mg PO qD) 14-21 days
  Other Names: Tarceva and Sprycel
  Arms: Arm C
Drug: Placebo — Placebo for 14-21 days.
  Arms: Arm D
Drug: Erlotinib — Erlotinib 150 mg for 14-21 days.
  Other Names: Tarceva
  Arms: Arm A

SUMMARY:
The central hypothesis to be tested in this study is that dual blockade of EGFR and Src pathways or proteins are distinct compared to inhibition of either kinase alone in head and neck and lung cancers.

DETAILED DESCRIPTION:
Background Head and neck squamous cell carcinoma (HNSCC) constitutes 3% of all malignancies and is the sixth most common malignancy worldwide. There will be an estimated 40,000 new cases and 11,000 deaths in the United States in 2007 and approximately 500,000 cases worldwide yearly [1]. Squamous cell carcinoma accounts for at least 90% of all head and neck cancers. Surgical resection remains a standard treatment for patients with resectable HNSCC. For patients with high risk of local or distant relapse, radiation therapy (RT) alone, or in combination with chemotherapy, is given after surgery to improve loco-regional control and overall survival. Moreover, surgery often represents the only curative option in patients who relapse locoregionally. Non-small cell lung cancer (NSCLC) is the leading cause of death worldwide. NSCLC is infrequently diagnosed when the cancer can be eradicated with surgical extirpation.

Specific Aims

* To determine the modulation of biomarkers by EGFR and/or Src targeting in head and neck and lung cancers.
* To determine if biomarker modulation is associated with reduction of tumor volume and/or evidence of histologic response in the tumor (e.g. decreased proliferation and/or decreased apoptosis) as well as safety and tolerability.

Subject population Patients will be accrued from head and neck and lung cancer patients who are surgical candidates. Surgery will be the primary curative treatment for patients enrolled in this study. Patients should not require any standard induction treatment prior to surgery. Surgery will have to be the best treatment option as determined by the treating physician. Therefore, we will not be delaying chemoradiotherapy or other curative treatment. We plan to include any stage of HNSCC or NSCLC that will be managed by primary surgery. If surgery is unexpectedly cancelled, the patient will be removed from the study unless there is an accessible lesion for biopsy. Ideally, the pre-treatment biopsy and the intraoperative sample will be obtained from the same site (when there are multiple lesions). Please see Section 3.0 for detailed eligibility criteria.

Treatment Plan The study drug or placebo will be taken for 14-21 days, and will be discontinued one day prior to planned surgical resection. If surgery is delayed, the study drug or placebo will be continued until one day prior to surgery, for up to a maximum of 28 days. Seven days is the minimum treatment for the patients to be evaluated. The interval between the last dose of experimental drug and surgery will be 12-36 hours. Please see Section 5.0 for treatment plan details. If the combination of erlotinib and dasatinib results in toxicity leading to a delay in surgery, the study will be terminated.

Statistical design and sample size This is a 4-arm randomized trial that is intended to estimate the effects of short-term preoperative therapy with EGFR and Src inhibitors upon a panel of biomarkers. The 4 treatment arms are erlotinib, dasatinib, their combination, and a placebo. We anticipate accruing 56 evaluable patients (14 patients per arm).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, head and neck or lung cancers
* Any NSCLC histology is eligible. Stages I, II, IIIA (T3N1 only) or recurrent NSCLC that will be managed with surgery are eligible.
* Primary tumors of any head and neck (oral cavity, oropharynx, hypopharynx, or larynx) or lung site will be included.
* Surgical resection of head and neck or lung must be planned, either as primary treatment or salvage. Patients must have tissue available prior to receiving drug(s).
* Age greater then 18 years.
* ECOG performance status 0-2.
* Women of childbearing potential (WOCBP) must have:

  1. A negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration
  2. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
  3. Ability to take oral medication (dasatinib must be swallowed whole).
  4. Concomitant Medications
* Patients agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib).
* Patient agrees that IV biphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
* Adequate hematologic, renal and hepatic function.
* Have signed written informed consent including a HIPPA form according to institutional guidelines.

Exclusion Criteria:

* Subjects who fail to meet the above criteria.
* Prior therapy for head and neck or lung cancers is allowed, with the exception of EGFR inhibitors. Any systemic therapy should have been completed at least 30 days prior to study enrollment.
* Pregnancy or breastfeeding. Women (patients or partners of male patients) of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy.
* Any unresolved chronic toxicity grade greater or equal to 2 from previous anticancer therapy (except alopecia and anemia).
* Acute hepatitis, known HIV, or active uncontrolled infection.
* Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment.
* Prior treatment with an EGFR inhibitor (tyrosine kinase inhibitor).
* Cardiac Symptoms; any of the following should be considered for exclusion:

  1. History of thromboembolic event or other condition currently requiring anticoagulation with warfarin (Coumadin). Patients whose therapy is changed to heparin is eligible.
  2. History of any other cancer except basal cell carcinoma of the skin.
  3. Concurrent medical condition which may increase the risk of toxicity, including:

     * Pleural or pericardial effusion of any grade
  4. History of significant bleeding disorder unrelated to cancer, including:

     * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
     * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
     * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding.
  5. Concomitant Medications, any of the following should be considered for exclusion:

     * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)
  6. Women who:

     * are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug,
     * have a positive pregnancy test at baseline, or
     * are pregnant or breastfeeding.
  7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are comprised of a panel of tumor proteins to be obtained before after administration of the study drugs. | 2-3 week preoperative period of drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Grandis, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Bauman JE, Duvvuri U, Gooding WE, Rath TJ, Gross ND, Song J, Jimeno A, Yarbrough WG, Johnson FM, Wang L, Chiosea S, Sen M, Kass J, Johnson JT, Ferris RL, Kim S, Hirsch FR, Ellison K, Flaherty JT, Mills GB, Grandis JR. Randomized, placebo-controlled window trial of EGFR, Src, or combined blockade in head and neck cancer. JCI Insight. 2017 Mar 23;2(6):e90449. doi: 10.1172/jci.insight.90449. PMID 28352657
- [Derived] Van Allen EM, Lui VW, Egloff AM, Goetz EM, Li H, Johnson JT, Duvvuri U, Bauman JE, Stransky N, Zeng Y, Gilbert BR, Pendleton KP, Wang L, Chiosea S, Sougnez C, Wagle N, Zhang F, Du Y, Close D, Johnston PA, McKenna A, Carter SL, Golub TR, Getz G, Mills GB, Garraway LA, Grandis JR. Genomic Correlate of Exceptional Erlotinib Response in Head and Neck Squamous Cell Carcinoma. JAMA Oncol. 2015 May;1(2):238-44. doi: 10.1001/jamaoncol.2015.34. PMID 26181029
- [Derived] Gross ND, Bauman JE, Gooding WE, Denq W, Thomas SM, Wang L, Chiosea S, Hood BL, Flint MS, Sun M, Conrads TP, Ferris RL, Johnson JT, Kim S, Argiris A, Wirth L, Nikiforova MN, Siegfried JM, Grandis JR. Erlotinib, erlotinib-sulindac versus placebo: a randomized, double-blind, placebo-controlled window trial in operable head and neck cancer. Clin Cancer Res. 2014 Jun 15;20(12):3289-98. doi: 10.1158/1078-0432.CCR-13-3360. Epub 2014 Apr 11. PMID 24727329